CLINICAL TRIAL: NCT03543423
Title: Studier af Den Tidlige Måltidsfase i Raske Individer
Brief Title: Studies of the Early Meal Phase in Healthy Individuals - Nutrient Absorption and Gastrointestinal Hormone Secretion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Simon Veedfald, Post doc, University of Copenhagen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UC/RH-early phase
Record Dates: First submitted 2018-05-20; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: Gut hormone secretion; Glucose absorption; early meal phase; Insulin and glucagon secretion
MeSH Terms: conditions — Insulin Resistance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Intervention Model Description: 12 healthy male individuals will each be studied on two occasions in random order.
  * oral glucose tolerance test
  * liquid mixed meal test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral glucose tolerance test (Experimental): Intervention: oral glucose tolerance test (75 gram glucose supplemented with 5g 3-OMG and 1g paracetamol) ingested over 2 min.
  Interventions: Other: Oral glucose tolerance test
- Liquid mixed meal test (Experimental): Intervention: Standardised liquid mixed meal (supplemented with 1g paracetamol) ingested over 2min
  Interventions: Other: Liquid mixed meal test

INTERVENTIONS:
Other: Oral glucose tolerance test — Oral glucose tolerance test will be carried out with a glucose solution made up of 75g glucose dissolved in 300mL. To the glucose solution will be added 5g 3-OMG and 1g paracetamol 5g 3-OMG
  Arms: Oral glucose tolerance test
Other: Liquid mixed meal test — A standardised liquid mixed meal test will be carried out using a standard liquid mixed meal (fresubin drink supplemented with 1g paracetamol).
  Arms: Liquid mixed meal test

SUMMARY:
To investigate gastrointestinal hormone secretions and nutrient absorption during the early meal phase we will recruit 12 healthy young men. They will be equipped with peripheral intravenous catheters for frequent blood sampling. Participants will be screened and acclimatised to the study situation on visit 1. On visit 2 and 3 participants will in random order ingest an oral glucose solution or a standardised liquid mixed meal over 2-3 min.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40years
* Male
* Normal Haemoglobin concentration
* Informed consent

Exclusion Criteria:

* Diabetes mellitus
* Family history of diabetes mellitus
* intestinal disease (for example inflammatory bowel disease or malabsorption)
* Family history of inflammatory bowel disease
* Previous intestinal resection (except uncomplicated appendicectomy)
* Body mass index (BMI) > 25 kg/m2
* Tobacco use
* kidney disease (se-creatinine> 130 µM and/or albuminuria)
* liver disease (ALAT and/or ASAT >2 × above normal range)
* Heart disease
* Treatment with drugs
* History of constipation
* Conditions with delayed or accelerated gastric emptying
* Latex or other allergies
* Bleeding diathesis

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasma GIP concentrations | -40, -20, -18, -16, -14, -12, -10, -8, -6, -4, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Glucose-dependent insulinotropic polypeptide plasma concentrations

SECONDARY OUTCOMES:
Plasma GLP-1 concentrations | -40, -20, -18, -16, -14, -12, -10, -8, -6, -4, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Glucagon-like peptide-1 plasma concentrations
Serum 3-OMG concentrations | -10, -2, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30
  Serum 3-OMG concentrations (glucose absorption marker)
Serum C-peptide and insulin concentrations | -40, -20, -18, -16, -14, -12, -10, -8, -6, -4, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Glucagon-like peptide-1 plasma concentrations
Plasma gastrin concentrations | -40, -20, -18, -16, -14, -12, -10, -8, -6, -4, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Plasma gastrin concentrations
Plasma CCK concentrations | -40, -20, -18, -16, -14, -12, -10, -8, -6, -4, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Plasma cholecystokinin concentrations
Plasma PP concentrations | -40, -20, -18, -16, -14, -12, -10, -8, -6, -4, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Plasma pancreatic polypeptide concentrations
Plasma NT concentrations | -40, -20, -18, -16, -14, -12, -10, -8, -6, -4, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Plasma Neurotensin concentrations
Plasma glucagon concentrations | -40, -20, -18, -16, -14, -12, -10, -8, -6, -4, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Plasma glucagon concentrations
Serum 3-OMG concentrations | -40, -20, -18, -16, -14, -12, -10, -8, -6, -4, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Serum 3-OMG concentrations (glucose absorption marker)
Plasma acetaminophen | -10, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Plasma acetaminophen (as a measure of gastric emptying)
Plasma amino acids | -10, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Plasma amino acids
Plasma bile acids | -10, -2, 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 30 min
  Plasma bile acids

CONTACTS AND LOCATIONS:
Overall Officials: Jens J Holst, DMSCI, Principal Investigator — Department of Biomedical Sciences
Locations (1):
- Department of Gastrointestinal Surgery, Righospitalet, Copenhagen, Capital, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Veedfald S, Rehfeld JF, van Hall G, Svendsen LB, Holst JJ. Entero-Pancreatic Hormone Secretion, Gastric Emptying, and Glucose Absorption After Frequently Sampled Meal Tests. J Clin Endocrinol Metab. 2022 Jan 1;107(1):e188-e204. doi: 10.1210/clinem/dgab610. PMID 34479362